CLINICAL TRIAL: NCT05249309
Title: Naturalistic Study of Ketamine in the Treatment of Depression: Suicide Risk Assessment and Serum Measurements of SIRT3, suPAR, hsCRP, Interleukin 6, Complete Blood Count, Leptin, Lipid Profile and Blood Glucose
Brief Title: Naturalistic Study of Ketamine in the Treatment of Depression
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Rio Grande do Sul (Other); Hospital Moinhos de Vento (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-0334
Record Dates: First submitted 2021-12-07; First posted 2022-02-21 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Major Depressive Disorder; Bipolar Disorder; Bipolar Depression; Bipolar I Disorder; Bipolar II Disorder; Affective Disorder
Keywords: Ketamine; Suicide; Depression; Major depressive disorder; Major depression; Unipolar depression; Depressive disorders; Bipolar I disorder; Bipolar II disorder; Bipolar depression
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder; Mood Disorders; Suicide; Depression; Depressive Disorder | interventions — Ketamine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — The types of biospecimens to be retained (plasma and serum).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treatment: The administration will be done subcutaneously, in the abdominal wall, using ketamine without dilution. The ketamine dose will be 0.5mg/kg, recommended for the first infusion. If there is no adequate response, according to psychiatric scales and clinical evaluation, the second infusion must be performed at least two days after the first, using 0.75mg/kg and the subsequent 1mg/kg. If the patient adequately responds to a dose (0.5 or 0.75mg/kg), it should be repeated after over twice weekly over a period of 4 weeks.
  Interventions: Drug: Ketamine
- Control: Will be checked weight, height and waist circumference and collected about 15 mL of peripheral blood.

INTERVENTIONS:
Drug: Ketamine — The administration will be done subcutaneously, in the abdominal wall, using ketamine without dilution. The ketamine dose will be 0.5mg/kg, recommended for the first infusion. If there is no adequate response, according to psychiatric scales and clinical evaluation, the second infusion must be performed at least two days after the first, using 0.75mg/kg and the subsequent 1mg/kg. If the patient adequately responds to a dose (0.5 or 0.75mg/kg), it should be repeated after over twice weekly over a period of 4 weeks.
  Other Names: Ketalar
  Groups: Treatment

SUMMARY:
This study aims to examine the effect of ketamine in decreasing the risk of suicide in patients with depression and its effectiveness as an antidepressant agent.

DETAILED DESCRIPTION:
Mood disorders are chronic, recurrent, and highly prevalent health conditions worldwide. Major depression and bipolar disorder are often associated with psychosocial functional impairments and general medical conditions. Furthermore, suicide figures as one of the most important negative outcomes of mood disorders. In this sense, according to the World Health Organization (WHO), psychiatric disorders are associated with more than 90% of cases of complete suicide and are responsible for 30% of reported suicide cases worldwide. Suicide is a matter of concern for clinicians, not only because of the individual and familiar impact but also due to its social and population impact; then, research involving new potential treatments for suicide behavior ate highly needed.

The literature has shown that ketamine, a substance commonly used as an anesthetic, is effective in treating depressive symptoms. Considering the high rate of suicide among patients with mood disorders and its consequences, the aim of this naturalistic study is to investigate the effect of ketamine in reducing the risk of suicide in patients with a depressive episode. The hypothesis is that treatment with ketamine will result in an improvement in depressive symptoms as well as in a decrease in the risk of suicide.

Therefore, forty-five patients will be recruited, with major depressive disorder, bipolar I disorder or bipolar II disorder and who were already on ketamine treatment prescribed by assistant psychiatrist (inclusion criteria). Patients will go on the standard protocol of ketamine 0.5mg/kg subcutaneously (SC) twice a week for one month in general. In line with a naturalistic approach, all changes in the protocol, in time and doses will be accepted, according to the assistant doctor prescription without study intervention.

After this period, they could receive the same dose of the medication once a week for the third month. In addition, patients will be monitored by phone until month six.

Forty-five participants without any personal or first-degree family history of psychiatry or neurologic disorders will be recruited to participate as controls. Biochemical analyses will be used to investigate inflammatory markers, transcription factors and other peripheral biomarkers in patients with mood disorders and healthy controls.

ELIGIBILITY:
Inclusion criteria

Having a diagnosis according to DSM-5 for

* Major depressive episode as part of either Major depressive disorder, Bipolar I disorder, or Bipolar II disorder according to Fifth Edition of Diagnostic and Statistical Manual for Mental Disorders (DSM-5);
* 18 years old or older;
* Be able to provide written informed consent.episode;
* MADRS scale total score ≥ 12 and score in items 1 (apparent sadness) and 2 (expressed sadness) ≥ 2 during the screening period (baseline);
* YMRS scale total score ≤ 11 at baseline;
* Having current symptoms of suicidal ideation and/or behavior, according to the C-SSRS scores;
* Use of effective contraceptive methods in the case of heterosexual women of childbearing age;
* Indication/prescription of the attending physician for the use of ketamine, subcutaneous;
* For the patients with Bipolar I disorder: currently using lithium, valproic acid, or atypical antipsychotic at therapeutic doses for at least four weeks prior to initial evaluation.
* For patients with Bipolar II disorder: currently using lithium, valproic acid, lamotrigine, or atypical antipsychotic at therapeutic doses for at least four weeks prior to initial evaluation.

Exclusion Criteria

* Patients with an unstable, defined, or suspected systemic medical condition;
* Women who are pregnant, breastfeeding or planning to become pregnant within the next year;
* Patients who cannot tolerate the use of ketamine or who have previous adverse effects associated with ketamine;
* Inability to comply with informed consent or treatment protocol needs;
* Patients currently with psychotic symptoms (according to DSM-5 criteria);
* Patients with a current diagnosis of any active substance use disorder according to the MINI/DSM-5 criteria (with the exception of tobacco);
* Patients with autoimmune or inflammatory conditions, cancer or active infectious diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Forty-five patients who fulfill the DSM-5 criteria for either MDD, Bipolar I disorder, or Bipolar II disorder who are currently in depressive episodes according to the structured clinical interview of the MINI. All participants must have been referred to receive ketamine for the treatment of a depressive episode at the Hospital de Clinicas de Porto Alegre (HCPA) and Hospital Moinhos de Vento (HMV).
  Forty-fiver participants without any personal or first-degree family history of psychiatry or neurologic disorders will be recruited to participate as controls. Biochemical analyses will be used to investigate inflammatory markers, transcription factors and other peripheral biomarkers in patients with mood disorders and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Changes in Columbia Suicide Severity Rating Scale (C-SSRS) - Ideation Severity | For Weeks 1, 2, 3, 4, 8, 12, 16, 20 and 24
  Intensity of ideation was measured using the C-SSRS for Suicide Ideation intensity of ideation item. Item responses range from 1 (wish to be dead) to 5 (active suicidal ideation with specific plan and intent), with higher scores indicating more severe ideation.
Changes in Columbia Suicide Severity Rating Scale (C-SSRS) - Behavior | For Weeks 1, 2, 3, 4, 8, 12, 16, 20 and 24
  Items measuring attempt behavior (number of Actual Attempts, number of Aborted Attempts, number of Interrupted Attempts) From the C-SSRS were summed to create a composite variable indexing attempt behavior. Higher scores indicate more attempt behavior.

SECONDARY OUTCOMES:
Change in depressive symptoms according to Hamilton Depression Rating Scale (HAMD) | For Weeks 1, 2, 3, 4, 8, 12, 16, 20 and 24
  Change from baseline in HAMD score. The 17-item HAMD measures depression severity. Each item was evaluated and scored using either a 5-point scale (e.g. absent, mild, moderate, severe, very severe) or a 3-point scale (e.g. absent, mild, marked). The total score of HAMD-17 may range from 0 (normal) to 52 (severe).
Change in psychotic symptoms according to Brief Psychiatric Rating Scale (BPRS) | For Weeks 1, 2, 3, 4, 8, 12, 16, 20 and 24
  Change from baseline in BPRS score. Scale range: from 0 to 108. Higher values represent more severe symptoms of psychosis.
Change in depressive symptoms according to Montgomery-Asberg Depression Rating Scale (MADRS) | For Weeks 1, 2, 3, 4, 8, 12, 16, 20 and 24
  MADRS is a 10-item rating scale for depressive mood symptoms severity, items rated on 0-6 scale, with total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms).
Change in remission of manic symptoms according to Young Mania Rating Scale (YMRS) | For Weeks 1, 2, 3, 4, 8, 12, 16, 20 and 24
  Change from baseline in YMRS score. The YMRS is a clinician-rated, 11-item checklist used to measure the severity of manic episodes. Information for assigning scores is gained from the participant's subjective reported symptoms over the previous 48 hours and from clinical observation during the interview. Seven items are ranked 0 through 4 and have descriptors associated with each severity level. Four items (irritability, speech, content, and disruptive-aggressive behavior) are scored 0 through 8 and have descriptors for every second increment. The total scale is 0-60. A score of ≤12 indicates remission of manic symptoms, and higher scores indicate greater severity of mania. Negative change from baseline scores indicate a decrease in severity of mania.
Change in functioning according to Functioning Assessment Short Test (FAST) | For Weeks 1, 2, 3, 4, 8, 12, 16, 20 and 24
  Change from baseline in FAST scores. The overall FAST score ranges from 0 to 72, where a higher score indicates more severe difficulties.
Change in SIRT3 levels in the blood. | For Weeks 1 and 4
  Change in Sirtuin 3 levels in the blood
Change in suPAR levels in the blood. | For Weeks 1 and 4
  Change in soluble urokinase-type plasminogen activator receptor levels in the blood
Change in hsCRP levels in the blood. | For Weeks 1 and 4
  Change in sensitivity C-reactive protein levels in the blood
Change in IL-6 levels in the blood. | For Weeks 1 and 4
  Change in interleukin 6 levels in the blood
Change in leptin levels in the blood. | For Weeks 1 and 4
  Change in leptin levels in the blood.
Change in blood count. | For Weeks 1 and 4
  Change in blood count.
Change in lipid profile levels in the blood. | For Weeks 1 and 4
  Change in lipid profile levels in the blood.
Change in blood glucose levels. | For Weeks 1 and 4
  Change in blood glucose levels.
Change in body weight | For Weeks 1 and 4
  The measurement of body weight will be carried out with individuals barefoot, wearing as little clothing as possible and positioned in the center of the platform while reading. Electronic scale with maximum capacity of 150 kg and precision of 0.1 kg.
  The weight will be measured in kilograms (kg).
Body height measurement | For Weeks 1 and 4
  The measurement of body height will be performed with barefoot individuals. The height will be measured in meters (m).
Change in the Body Mass Index (BMI) | For Weeks 1 and 4
  Weight and height will be combined to report BMI in kg/m^2.
Change in waist circumference | For Weeks 1 and 4
  The waist circumference (WC) will be measured with the aid of an inelastic measuring tape of 1.5 m in length and 0.1 cm accuracy. The measurement will be taken with the patient standing, in upright position, relaxed abdomen, arms extended along the body and feet apart in a distance of 25-30 cm. The midpoint between the iliac crest and the lower edge of the last rib, standing upright, with no clothes on the chest and at the end of expiration.
Change in blood pressure | For Weeks 1, 2, 3 and 4
  Change in diastolic and systolic blood pressure during ketamine application
Change in IL-10 levels in the blood. | For Weeks 1 and 4
  Change in interleukin 10 levels in the blood
Change in TNFalpha levels in the blood. | For Weeks 1 and 4
  Change in TNFalpha levels in the blood
Change in the Dietary Inflammatory Index (DII) | For Weeks 1 and 4
  The inflammatory index of the diet will be calculated from the average of dietary recalls in the last 24 hours (R24h) at the interview with intervals between them according to the application of ketamine.
  A high DII score reflects pro-inflammatory potential of the diet, whereas a low DII score reflects the anti-inflammatory potential of the diet.
Changes in proteomic markers | For Weeks 1 and 4
  Proteomic markers will be analyzed at weeks 1 and 4 to observe for any treatment-emergent changes to increase the predictive validity of the proteomic signatures.

CONTACTS AND LOCATIONS:
Overall Officials: Ana P Anzolin, Master, Study Chair — Laboratory of Molecular Psychiatry, Hospital de Clínicas de Porto Alegre; Keila Maria M Ceresér, PhD, Study Chair — Laboratory of Molecular Psychiatry, Hospital de Clínicas de Porto Alegre; Jéferson F Goularte, PhD, Study Chair — Laboratory of Molecular Psychiatry, Hospital de Clínicas de Porto Alegre; Jairo Vinícius Pinto, MD, PhD, Study Chair — Laboratory of Molecular Psychiatry, Hospital de Clínicas de Porto Alegre; Paulo B de Abreu, MD, PhD, Study Director — Laboratory of Molecular Psychiatry, Hospital de Clínicas de Porto Alegre; Ives C Passos, MD, PhD, Study Chair — Laboratory of Molecular Psychiatry, Hospital de Clínicas de Porto Alegre; Márcia K Sant'Anna, MD, PhD, Principal Investigator — Laboratory of Molecular Psychiatry, Hospital de Clínicas de Porto Alegre; Ellen Scotton, Master, Study Chair — Laboratory of Molecular Psychiatry, Hospital de Clínicas de Porto Alegre; Luciane N Cruz, MD, PhD, Study Director — Hospital Moinhos de Vento
Locations (2):
- Brazil (2):
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cordova VHS, Anzolin AP, Sant'Ana MK, Lacerda A, Belmonte-de-Abreu PS. Allergic reaction induced by subcutaneous administration of ketamine: a case report. Int Clin Psychopharmacol. 2022 Sep 1;37(5):229-230. doi: 10.1097/YIC.0000000000000411. Epub 2022 May 2. PMID 35503059
- [Derived] Anzolin AP, Baldez DP, Montezano BB, Kapczinski F, de Abreu PB, Kauer-Sant'Anna M. Subcutaneous ketamine reduces suicide risk and improves functioning in depression: A proof-of-concept study. Psychiatry Res. 2024 Jul;337:115915. doi: 10.1016/j.psychres.2024.115915. Epub 2024 Apr 20. PMID 38688118
- [Derived] Anzolin AP, Goularte JF, Pinto JV, Belmonte-de-Abreu P, Cruz LN, Cordova VHS, Magalhaes LS, Rosa AR, Cereser KM, Kauer-Sant'Anna M. Ketamine study: Protocol for naturalistic prospective multicenter study on subcutaneous ketamine infusion in depressed patients with active suicidal ideation. Front Psychiatry. 2023 Mar 9;14:1147298. doi: 10.3389/fpsyt.2023.1147298. eCollection 2023. PMID 36970275